CLINICAL TRIAL: NCT05398029
Title: Open-label, Phase 1b, Single-ascending Dose and Optional re Dosing Study to Evaluate the Safety of VERVE-101 Administered to Patients With Heterozygous Familial Hypercholesterolemia, Atherosclerotic Cardiovascular Disease, and Uncontrolled Hypercholesterolemia
Brief Title: A Study of VERVE-101 in Patients With Familial Hypercholesterolemia and Cardiovascular Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verve Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VT-1001
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Heterozygous Familial Hypercholesterolemia; Atherosclerotic Cardiovascular Disease; Hypercholesterolemia
Keywords: VERVE-101; Familial Hypercholesterolemia; Cardiovascular Disease; Dose Escalation; Gene Editing; Base Editing
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Hyperlipoproteinemia Type II; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single ascending dose escalation/adaptive design followed by single dose expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A: Single Ascending Dose Escalation/Adaptive Design (Experimental): Participants will receive a single dose of VERVE-101 in multiple dose-escalation cohorts.
  Interventions: Drug: VERVE-101
- Part B: Single Dose Expansion (Experimental): Participants will receive a single dose of VERVE-101 selected based on the doses studied in Part A.
  Interventions: Drug: VERVE-101

INTERVENTIONS:
Drug: VERVE-101 — Intravenous (IV) infusion.

SUMMARY:
VT-1001 is an open-label, phase 1b, single-ascending dose study that will evaluate the safety of VERVE-101 administered to patients with heterozygous familial hypercholesterolemia (HeFH), atherosclerotic cardiovascular disease (ASCVD), and uncontrolled hypercholesterolemia. VERVE-101 uses base-editing technology designed to disrupt the expression of the PCSK9 gene in the liver and lower circulating PCSK9 and LDL-C in patients with established ASCVD due to HeFH. This study is designed to determine the safety and pharmacodynamic profile of VERVE-101 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female participants 18 up to 75 years at time of signing of informed consent
* Female participants not of child-bearing potential
* Diagnosis of HeFH
* Established ASCVD

Exclusion Criteria:

* Active or history of chronic liver disease
* Current treatment with PCSK9 monoclonal antibody therapy
* Current or past treatment with inclisiran
* Clinically significant or abnormal laboratory values as defined by the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs). | up to Day 365

SECONDARY OUTCOMES:
Evaluation of maximum observed concentration (Cmax) | up to Day 365
Evaluation of time to maximum observed concentration (tmax) | up to Day 365
Evaluation of terminal elimination half-life (t1/2) | up to Day 365

OTHER OUTCOMES:
Percent and absolute change from baseline in plasma PCSK9 concentration. | up to Day 365
Percent and absolute change from baseline in LDL-C. | up to Day 365

CONTACTS AND LOCATIONS:
Locations (3):
- New Zealand (2):
  - Clinical Study Center, Auckland
  - Clinical Study Center, Christchurch
- Clinical Study Center, London, United Kingdom